CLINICAL TRIAL: NCT06252584
Title: Multi-peptide Vaccination Adjuvanted With the TLR1/2 Ligand XS15 in Acute Myeloid Leukemia (AML) Patients Who Have Achieved Complete Remission With First Line Therapy
Brief Title: Multi-peptide Vaccination Adjuvanted With XS15 in Acute Myeloid Leukemia Patients
Acronym: AML-VAC-XS15
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AML-VAC-XS15-01
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-01

CONDITIONS: Acute Myeloid Leukemia, Adult
Keywords: acute myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Protein Subunit Vaccines

STUDY DESIGN:
Intervention Model Description: Single Arm Treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multipeptide Vaccination (Experimental): The vaccine cocktail will be administered subcutaneously (s.c.) together with the TLR1/2 ligand XS15 (50 μg) emulsified in Montanide ISA 51 VG (1:1) as adjuvant. Two vaccinations within a 6-week interval are planned, with the option of one additional booster in case of insufficient response after the first two vaccinations. Peptide vaccination will take place in AML patients that have achieved a morphological complete remission (CR) or a complete remission with incomplete blood count recovery (CRi) with standard first line treatment. MRD positivity is permitted. Vaccination will start 4-28 weeks after last application of intensive chemotherapy). Any maintenance treatment, e.g. with oral azacytidine or midostaurin, or ongoing low intensity therapy, e.g. with HMA, venetoclax etc. is permitted, can be applied throughout the vaccination and continued after study treatment according to the treating physician's decision.
  Interventions: Drug: Vaccines, Peptide

INTERVENTIONS:
Drug: Vaccines, Peptide — Multi-peptide vaccine cocktail comprising 9 different immunopeptidome-defined mutated and non-mutated AML/ leukemia stem and progenitor cell (LSC)-associated HLA class I and HLA class II peptides. The vaccine cocktail is synthesized and formulated in the GMP-certified Wirkstoffpeptidlabor at the University of Tübingen.
  Other Names: Multipeptide Vaccine AML-VAC-XS15

SUMMARY:
The aim of this Phase I study is to evaluate the immunogenicity along with safety and toxicity as well as first efficacy of a multi-peptide vaccine adjuvanted with the TLR1/2 ligand XS15 emulsified in Montanide ISA 51 VG (AML-VAC-XS15) in AML patients who have achieved CR or CRi with first line treatment.

DETAILED DESCRIPTION:
Peptide vaccine: Multi-peptide vaccine cocktail comprising 9 different immunopeptidome-defined mutated and non-mutated AML/ leukemia stem and progenitor cell (LSC)-associated HLA class I and HLA class II peptides.

The vaccine cocktail is synthesized and formulated in the GMP-certified Wirkstoffpeptidlabor at the University of Tübingen (headed by Juliane Walz).

Treatment schedule:

The vaccine cocktail will be administered subcutaneously (s.c.) together with the (toll-like receptor )TLR1/2 ligand XS15 (50 µg) emulsified in Montanide ISA 51 VG (1:1) as adjuvant.

Two vaccinations within a 6-week interval are planned, with the option of one additional booster in case of insufficient response after the first two vaccinations.

Peptide vaccination will take place in AML patients that have achieved a morphological complete remission (CR) or a complete remission with incomplete blood count recovery (CRi) with standard first line treatment. Minimal residual disease (MRD) positivity is permitted.

Vaccination will start 4-28 weeks after last application of intensive chemotherapy). Any maintenance treatment, e.g. with oral azacytidine or midostaurin, or ongoing low intensity therapy, e.g. with HMA, venetoclax etc. is permitted, can be applied throughout the vaccination and continued after study treatment according to the treating physician's decision.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged ≥18 years of age
* Existence of a written informed consent
* Documented diagnosis of AML according to WHO guidelines

  * morphological complete remission (CR) or complete remission with incomplete blood count recovery (CRi)
  * positive MRD is permitted
  * completion of previous intensive therapy (first vaccination 4-28 weeks after last application of chemotherapy) or
  * ongoing low intensity treatment with e.g. hypomethylating agents (HMA), venetoclax, etc.
  * ongoing maintenance treatment with e.g. oral azacytidine or midostaurin is permitted.
  * not eligible for allogeneic stem cell transplantation
* Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 2
* Adequate organ function laboratory values.

  * bilirubin ≤ 3 times upper limit range (exception isolated indirect hyperbilirubinemia (Morbus Gilbert-Meulengracht)).
  * alanine aminotransferase (ALT) and aminotransferase (AST), ≤ 5 times upper limit range
  * creatinine clearance GFR > 30 ml/min (CKD-EPI)
  * platelets > 50.000/μl
  * absolute CD3+ T cell count ≥ 200/μl
* negative serological hepatitis B test or negative PCR in case of positive serological test without evidence of an active infection, negative testing of hepatitis C RNA, negative HIV test within 6 weeks prior to study inclusion
* Female patients of child bearing potential (FCBP) and male patients with partners of child bearing potential, who are sexually active, must agree to the use of two effective forms (at least one highly effective method) of contraception (for more detailed information see chapter 5.7 Contraception, pregnancy, sperm donation and nursing). This should be started from the signing of the informed consent and be continued until 3 months (both female and male patients) after last vaccination).
* For FCBP two negative pregnancy tests (sensitivity of at least 25 mlU/mL) prior to first application of first vaccination, one at screening and the other prior (< 24 h) to first vaccination
* Postmenopausal or evidence of non-child-bearing status

Exclusion Criteria:

* Pregnant or breastfeeding.
* Unwilling or unable to follow the study schedule for any reason.
* Chemotherapy or other systemic therapy or radiotherapy, up to 14 days prior to the first dose of study drug (ongoing maintenance treatment or low intensity treatment is permitted).
* Concurrent or previous treatment within 28 days in another interventional clinical trial with an investigational anticancer therapy or any other investigational therapy, which would interfere with the study's primary and secondary endpoints.
* Major surgery within 28 days of dosing of study drug.
* Treatment with immunotherapy agents within 28 days of dosing of study drug.
* Diagnosis of acute promyelocytic leukemia (APL)
* Autoimmune disease that requires or has required treatment with systemic immunosuppressive treatments, except low dose corticosteroids (< 10 mg/ day), in the past 1 year.
* Prior history of malignancies, other than AML/myelodysplastic syndrome (MDS), unless the subject has been free of the disease for

  ≥ 2 years. Exceptions include the following: basal cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the breast, histological finding of prostate cancer of TNM stage T1
* Prior stem cell allograft or organ transplantation
* Ongoing or active infection (including SARS-CoV-2)
* Have received any live vaccination within 28 days prior to the first dose of AML-VAC-XS15.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-02 (Estimated); Primary Completion 2026-05-02 (Estimated); Study Completion 2026-11-02 (Estimated)

PRIMARY OUTCOMES:
immunogenicity | Visit 1( Day 0); Visit 2 (Day 42); End of Treatment (Day 70); Follow-Up (Day160); Follow-Up 1(Day 188); Follow-Up 2 (Day 250)
  Blood will be taken before peptide vaccination and during vaccination phase and follow-ups at each visit
  IFN-gamma ELISPOT Counts
  Percentage of patients with induction of an AML-VAC-XS15-specific specific T-cell response until End of study visit (EOS) compared to baseline as determined by IFNγ ELISPOT.